CLINICAL TRIAL: NCT00872300
Title: An Exploratory Phase II Study of PHA-739358 in Patients With Multiple Myeloma Harbouring the t(4;14) Translocation With or Without FGFR3 Expression
Brief Title: PHA-739358 for the Treatment of Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Nerviano Medical Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AURA-6202-011
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — danusertib

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: PHA-739358

INTERVENTIONS:
Drug: PHA-739358 — Weekly IV infusion for 3 consecutive weeks in a 4-week cycle

SUMMARY:
The purpose of this study is to determine the antitumor activity of PHA-739358 as single agent IV infusion in adult patients with Multiple Myeloma who have a history of at least 2 previous lines of treatment for the disease.

ELIGIBILITY:
Inclusion Criteria:

* active multiple myeloma progressing after at least 2 prior lines of treatment
* measurable disease
* t(4;14) translocation
* life expectancy of at least 3 months

Exclusion Criteria:

* uncontrolled hypertension
* myocardial infarction, unstable angina, symptomatic congestive heart failure, cerebrovascular accident in the past 6 months.
* pregnancy or breast feeding
* active infections, including HIV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-10; Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Response Rate according to International Myeloma Working Group uniform response criteria for multiple myeloma. | At end of each cycle

SECONDARY OUTCOMES:
Overall safety profile | All cycles

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - MAYO Clinic, Scottsdale, Arizona
  - The Robert H Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
- France (2):
  - Hôpital Huriez, Centre Hospitalier Régional Universitaire de Lille, Lille
  - University Hospital Hôtel-Dieu, Nantes